CLINICAL TRIAL: NCT01264575
Title: ED50 and ED95 of Intrathecal Bupivacaine With or Without Epinephrine for Total Knee Replacement Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul Medical Center (Other)
Responsible Party: Principal Investigator, Won Ho Kim, Staff Anesthesiologist, Seoul Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: SMC-2010-12-18
Record Dates: First submitted 2010-12-20; First posted 2010-12-22 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Spinal Anesthesia; Total Knee Replacement Arthroplasty
Keywords: spinal anesthesia; intrathecal bupivacaine; epinephrine; ED50; ED95
MeSH Terms: interventions — Epinephrine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (12):
- BPV6E1 (Experimental)
  Interventions: Drug: intrathecal bupivacaine 6 mg with 100 mcg of epinephrine
- BPV7E1 (Experimental)
  Interventions: Drug: intrathecal bupivacaine 7 mg with 100 mcg of epinephrine
- BPV8E1 (Experimental)
  Interventions: Drug: intrathecal bupivacaine 8 mg with 100 mcg of epinephrine
- BPV9E1 (Experimental)
  Interventions: Drug: intrathecal bupivacaine 9 mg with 100 mcg of epinephrine
- BPV10E1 (Experimental)
  Interventions: Drug: intrathecal bupivacaine 10 mg with 100 mcg of epinephrine
- BPV11E1 (Experimental)
  Interventions: Drug: intrathecal bupivacaine 11 mg with epinephrine 100 mcg
- BPV6E2 (Experimental)
  Interventions: Drug: intrathecal bupivacaine 6 mg with 200 mcg of epinephrine
- BPV7E2 (Experimental)
  Interventions: Drug: intrathecal bupivacaine 7 mg with 200 mcg of epinephrine
- BPV8E2 (Experimental)
  Interventions: Drug: intrathecal bupivacaine 8 mg with 200 mcg of epinephrine
- BPV9E2 (Experimental)
  Interventions: Drug: intrathecal bupivacaine 9 mg with 200 mcg of epinephrine
- BPV10E2 (Experimental)
  Interventions: Drug: intrathecal bupivacaine 10 mg with 200 mcg of epinephrine
- BPV11E2 (Experimental)
  Interventions: Drug: intrathecal bupivacaine 11 mg with 200 mcg of epinephrine

INTERVENTIONS:
Drug: intrathecal bupivacaine 6 mg with 100 mcg of epinephrine — intrathecal bupivacaine 6 mg with 100 mcg of epinephrine
  Other Names: marcaine; epinephrine
  Arms: BPV6E1
Drug: intrathecal bupivacaine 7 mg with 100 mcg of epinephrine — intrathecal bupivacaine 7 mg with 100 mcg of epinephrine
  Other Names: marcaine; epinephrine
  Arms: BPV7E1
Drug: intrathecal bupivacaine 8 mg with 100 mcg of epinephrine — intrathecal bupivacaine 8 mg with 100 mcg of epinephrine
  Other Names: marcaine; epinephrine
  Arms: BPV8E1
Drug: intrathecal bupivacaine 9 mg with 100 mcg of epinephrine — intrathecal bupivacaine 9 mg with 100 mcg of epinephrine
  Other Names: marcaine; epinephrine
  Arms: BPV9E1
Drug: intrathecal bupivacaine 10 mg with 100 mcg of epinephrine — intrathecal bupivacaine 10 mg with 100 mcg of epinephrine
  Other Names: marcaine; epinephrine
  Arms: BPV10E1
Drug: intrathecal bupivacaine 11 mg with epinephrine 100 mcg — intrathecal bupivacaine 11 mg with epinephrine 100 mcg
  Other Names: marcaine; epinephrine
  Arms: BPV11E1
Drug: intrathecal bupivacaine 6 mg with 200 mcg of epinephrine — intrathecal bupivacaine 6 mg with 200 mcg of epinephrine
  Other Names: bupivacaine; epinephrine
  Arms: BPV6E2
Drug: intrathecal bupivacaine 7 mg with 200 mcg of epinephrine — intrathecal bupivacaine 7 mg with 200 mcg of epinephrine
  Other Names: bupivacaine; epinephrine
  Arms: BPV7E2
Drug: intrathecal bupivacaine 8 mg with 200 mcg of epinephrine — intrathecal bupivacaine 8 mg with 200 mcg of epinephrine
  Other Names: bupivacaine; epinephrine
  Arms: BPV8E2
Drug: intrathecal bupivacaine 9 mg with 200 mcg of epinephrine — intrathecal bupivacaine 9 mg with 200 mcg of epinephrine
  Other Names: bupivacaine; epinephrine
  Arms: BPV9E2
Drug: intrathecal bupivacaine 10 mg with 200 mcg of epinephrine — intrathecal bupivacaine 10 mg with 200 mcg of epinephrine
  Other Names: bupivacaine; epinephrine
  Arms: BPV10E2
Drug: intrathecal bupivacaine 11 mg with 200 mcg of epinephrine — intrathecal bupivacaine 11 mg with 200 mcg of epinephrine
  Other Names: bupivacaine; epinephrine
  Arms: BPV11E2

SUMMARY:
This prospective randomized double-blind dose-response study is aimed to investigate the ED50 and ED95 of intrathecal bupivacaine with or without epinephrine 100 mcg for total knee replacement arthroplasty.

DETAILED DESCRIPTION:
Patients undergoing total knee replacement arthroplasty are randomly assigned to six bupivacaine dose group (6, 7, 8, 9, 10, 11 mg). Combined spinal-epidural anesthesia would be performed. The dose would be considered as successful if no epidural supplement was required during surgery. A probit analysis will be performed to calculate the ED50 and ED95 of intrathecal bupivacaine with or without epinephrine for total knee replacement arthroplasty.

After these measurements, ED50 and ED95 of bupivacaine with epinephrine would be compared with those without epinephrine.

ELIGIBILITY:
Inclusion Criteria:

* The patients with ASA class I or II scheduled for total knee replacement surgery

Exclusion Criteria:

* Patients with previous spine surgery, diabetic and other neuropathy, skin infection at the site of injection, allergy to bupivacaine and other common contraindications for spinal anesthesia were excluded from this study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2009-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
the success of anesthesia | during the surgery (average two hours)
  The individual dose would be considered to be successful if no epidural supplement is required during surgery.

SECONDARY OUTCOMES:
Adverse effects of the various intrathecal bupivacaine dose | during surgery (average two hours)
  lowest systolic blood pressure, vasopressure requirements, nausea, vomitting

CONTACTS AND LOCATIONS:
Overall Officials: Won Ho Kim, M.D., Principal Investigator — Seoul Medical Center
Locations (1):
- Seoul Medical Center, Seoul, South Korea